CLINICAL TRIAL: NCT07195786
Title: Expansion-floating Craniotomy for the Treatment of Malignant Cerebral Edema Caused by Acute Ischemic Stroke--A Prospective, Multicenter, Non-inferiority,Cohort Study（ECAIS）
Brief Title: Expansion-floating Craniotomy for the Treatment of Malignant Cerebral Edema Caused by Acute Ischemic Stroke
Acronym: ECAIS
Status: Not yet recruiting | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-230
Record Dates: First submitted 2025-09-15; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke, Acute; Malignant Cerebral Edema
Keywords: Expansion-floating Craniotomy; Malignant Cerebral Edema; decompressive craniectomy; Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Decompressive Craniectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Treatment group: Expansion-floating Craniotomy (EC) is performed, preserving the bone flap, while suspending it above the skull using specific fixation devices.
  Interventions: Procedure: Expansion-floating Craniotomy
- Standard treatment control group: Decompressive Craniectomy (DC) is performed, removing a section of skull bone to reduce intracranial pressure (ICP).
  Interventions: Procedure: decompressive craniectomy
- Conservative treatment group: Conservative pharmacological therapy was administered instead, as surgical intervention indicated per guidelines was refused by the patient or family.
  Interventions: Drug: drug conservative therapeutic

INTERVENTIONS:
Procedure: Expansion-floating Craniotomy — Following craniotomy with bone flap removal, cerebral edema is assessed. The bone flap is then elevated using 2-3 titanium connectors. The elevation height must be sufficient to at least prevent contact between the bone flap and the underlying brain tissue. If cerebral swelling proves less severe than anticipated or begins to subside, the connectors can be loosened minimally invasively after a maximum scalp expansion period of 7-10 days. The elevated bone flap gradually repositions itself. Mild compression is applied using an elastic bandage for fixation, thereby restoring cranial integrity.
  Groups: Treatment group
Procedure: decompressive craniectomy — The patient is placed supine with the head rotated contralaterally. A large retroauricular question-mark incision is made in the scalp. Alternatively, a Kempe incision or preauricular incision may be used according to surgeon preference. Meticulous preservation of the superficial temporal artery (STA) is essential during the procedure to prevent ischemic complications in the flap. After elevating the myocutaneous flap to expose the operative field, a fronto-temporo-parietal craniectomy is performed. For unilateral decompressive craniectomy, the bone window should measure at least 15 × 12 cm, extending inferiorly to the floor of the temporal fossa to ensure adequate decompression.
  Groups: Standard treatment control group
Drug: drug conservative therapeutic — Pharmacotherapy for malignant cerebral edema has been implemented according to current guidelines.
  Groups: Conservative treatment group

SUMMARY:
This clinical study investigates Expansion-floating Craniotomy (EC), a novel surgical technique for treating life-threatening malignant cerebral edema following large hemispheric infarction (commonly known as massive stroke). Malignant edema causes rapid increases in intracranial pressure, compressing vital brain structures and risking fatal brain herniation, requiring urgent intervention.

The current international standard treatment is traditional decompressive craniectomy (DC). DC involves removing a section of the skull to allow brain swelling, effectively reducing pressure and mortality risk. It is strongly recommended (Class I, Level A evidence) in major guidelines. However, DC typically requires a second major surgery (cranioplasty) approximately 3 months later to replace the removed bone flap, involving additional costs and risks like progressive intracranial hemorrhage or subdural hygroma.

EC is a newer approach designed to potentially eliminate the need for a second surgery. During EC, surgeons use medical titanium plates to temporarily elevate the bone flap, creating immediate space for brain swelling while keeping the bone flap attached. Once brain swelling subsides (usually within weeks), a minor procedure flattens the titanium plates, allowing the patient's own bone to naturally reposition without requiring cranioplasty. EC may be performed based on surgeon assessment of brain swelling, guideline considerations, or experience. If EC is deemed unsuitable during surgery, DC will be performed instead.

While early research suggests EC achieves decompression similar to DC while preserving the bone flap, its safety and effectiveness compared to the established DC procedure are not yet fully proven. DC is a well-understood, mature technique with known risks and benefits, including the certainty of needing cranioplasty. Conservative management is reserved for patients unfit for surgery but may not prevent neurological deterioration.This study aims to conduct a preliminary assessment of the outcomes of EC versus DC.

DETAILED DESCRIPTION:
Extensive cerebral infarction leads to progressive brain edema within 24-48 hours of ischemic injury. This edema can cause secondary damage over subsequent days through elevated intracranial pressure (ICP) and brain herniation. When edema is severe enough to cause decompensated ICP elevation, it is termed malignant edema, which can compromise potentially salvageable peri-infarct penumbral tissue.

Decompressive craniectomy (DC) is widely used to alleviate elevated ICP and prevent herniation. Cochrane reviews incorporating data from three major randomized trials (DECIMAL, DESTINY, HAMLET) demonstrate that DC improves survival and favorable outcomes compared to medical management alone. However, morbidity associated with DC and subsequent cranioplasty is significant, reaching up to 40%. Complications include delayed postoperative seizures (reported in 37-61.1% of cases), hydrocephalus (40%), neurological deficits like the syndrome of the trephined (26%), and chronic headaches often resolving only after cranioplasty (17%). Specific complication rates reported by Ban et al. include contralateral hematoma (5.6%), contusion expansion (12.4%), postoperative seizures (3.4%), external brain herniation (14.6%), CSF leakage (2.2%), infection (4.5%), subdural hygroma (32.6%), post-traumatic hydrocephalus (11.2%), and syndrome of the trephined (9.0%).

To address the limitations of DC, techniques like decompressive cranioplasty (DCP), also known as hinge craniotomy (HC), have been proposed. Unlike DC, HC preserves the bone flap, suspending it above the skull using specific fixation devices to avoid the long-term sequelae of bone removal. HC aims to reduce elevated ICP, prevent worsening edema and herniation, reduce the complexity of subsequent cranioplasty, and offer potential cost benefits. First described in 2007 for refractory post-traumatic ICP, HC has been used off-label for other indications. Potential advantages over DC include controlling moderate edema while avoiding a second major cranioplasty surgery, a crucial factor in resource-limited settings, and potentially lower complication rates.

However, HC may have limitations, primarily concerning the adequacy of the achieved expansion volume and potential subsequent need for conversion to DC. Early HC techniques reportedly provided only 40-60ml of expansion, potentially insufficient for malignant edema, though recent modifications claim volumes of 100-120ml. While some studies suggest comparable ICP control between HC and DC, rigorous data on HC's safety and efficacy, particularly its ability to sufficiently mitigate midline shift, brain swelling, and prevent herniation in large hemispheric infarctions, remain limited and require validation through systematic clinical studies.

Our team recently reported a novel technique termed Expansion-floating Craniotomy (EC). EC utilizes three peptide plates to elevate the bone flap to a predetermined position, ensuring adequate decompression while preserving the potential for outward displacement. As cerebral swelling subsides, subsequent loosening of the plates allows the bone flap to spontaneously reposition. EC was successfully implemented in four emergency cases, achieving the desired decompression volume while preserving the bone flap. This technique aims to provide optimal decompression without bone removal, potentially reducing complications associated with prior techniques. Potential advantages include superior cosmetic outcomes, maintenance of appropriate ICP, cost reduction, and simplified bone flap repositioning.

Study Design: This is a multicenter, non-inferiority cohort study. Patients with acute, large anterior circulation ischemic stroke will be allocated to one of three groups based on family consent:

Expansion-floating Craniotomy (EC) Group Decompressive Craniectomy (DC) Group Conservative Management Group

Objectives:

To evaluate the non-inferiority of EC compared to DC in treating patients with acute large anterior circulation infarction.

To further explore the clinical acceptability of the EC technique.

To assess differences in the postoperative complication profile, including:

Delayed intracranial hemorrhage (confirmed by CT >72 hours post-op) Incisional infection / CSF leakage rate Incidence of paradoxical brain herniation

ELIGIBILITY:
Inclusion Criteria:

* Age requirement: Adults aged >18 but <80 years
* Acute cerebral infarction diagnosis: Patients with internal carotid artery or middle cerebral artery occlusion within 48 hours, meeting all three criteria:

NIHSS score ≥16 with item 1a (level of consciousness) ≥1 CT demonstrating >50% MCA territory infarction or hypoperfused area >2/3, OR DWI hyperintensity volume >82 ml within 6 hours of onset, OR DWI infarct volume >145 ml within 14 hours

* Imaging evidence: Midline shift ≥5 mm to the contralateral side on CT, OR significant ipsilateral ventricular compression with effacement of cerebral sulci/cisterns.

Exclusion Criteria:

* Pre-stroke mRS score ≥1
* Significant contralateral cerebral infarction
* Symptomatic intracranial hemorrhage
* Any known coagulopathy
* Life expectancy <3 years
* Any severe comorbidities potentially interfering with treatment evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects developing malignant cerebral edema after acute cerebral infarction
Sampling Method: Non-Probability Sample
Enrollment: 356 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Functional outcomes assessed by the modified Rankin Scale (mRS) were dichotomized into scores 0-4 versus 5 and 6 | 3 months

SECONDARY OUTCOMES:
Median survival time | 3 months
  Median survival time (estimated by Kaplan-Meier method, from enrollment to death from any cause)
Overall mortality | 3 months
  Overall mortality（death from any cause）
Time interval from initial surgery to bone flap reimplantation or Expansion-Suspension Technique fixation (if applicable) | 3 months
Incidence of procedure-related complications | 3 months
  occurring after initial surgery or bone flap reimplantation, including: Transfusion-requiring surgical hemorrhage Anesthesia-related adverse events Pharmacologically-managed pain Impaired wound healing or surgical site infection Cerebrospinal fluid (CSF) leakage Abscess formation Any secondary complications prolonging hospitalization or requiring readmission (e.g., thrombosis, systemic infection, embolism
The Short-From-36 Health Survey（SF-36） | 3 months
  The SF-36 can be self-administered, completed by others, or conducted via telephone interview. The assessment typically takes 5 to 10 minutes, though it may require up to 15 minutes for older adults. Scoring involves calculating the sum of item scores across each subscale, weighted according to specific criteria, to obtain a raw subscale score. This raw score is then converted into a standardized score ranging from 0 to 100. Higher scores indicate better quality of life.
Hamilton Depression Scale | 3 months
  The Hamilton Depression Rating Scale is an observer-rated measure. Trained raters assess patients' symptoms and assign scores accordingly. It effectively reflects the severity of depression: milder symptoms correspond to lower total scores, while more severe symptoms result in higher total scores.We use 24-item version: Total score ≥35 points may indicate severe depression; Total score ≥20 points may indicate mild or moderate depression; Total score ≤8 points may indicate no depressive symptoms.
Barthel Index | 3 months
  Total Score Range: 0-100 points. Higher scores indicate greater self-care ability.
  Level Classification:
  Heavily Dependent: Total score ≤ 40 points. Requires comprehensive nursing care.
  Moderately Dependent: 41-60 points. Requires assistance for most activities. Mildly Dependent: 61-99 points. Requires minimal assistance. Independent: 100 points. Fully self-sufficient. Higher scores indicate better functional ability.

IPD SHARING:
Plan to Share IPD: No